CLINICAL TRIAL: NCT06410833
Title: Effectiveness of Belimumab After Rituximab in Resistant Primary Juvenile Sjogren's Syndrome
Brief Title: Belimumab After Rituximab in Resistant Primary Juvenile SS
Acronym: BRRPJS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Central South University (Other); Shenzhen Children's Hospital (Other Government); The First Hospital of Jilin University (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); The Affiliated Hospital of Qingdao University (Other); Children's Hospital of Nanjing Medical University (Other); Children's Hospital of Fudan University (Other); Shengjing Hospital (Other); Shanghai Children's Hospital (Other); Tianjin Children's Hospital (Other)
Responsible Party: Principal Investigator, Hongmei Song, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: K3926
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sjogren's Syndrome; Pediatric ALL
Keywords: Rituximab; Belimumab
MeSH Terms: conditions — Sjogren's Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Rituximab; belimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sequential use of rituximab and belimumab (Experimental)
  Interventions: Drug: Rituximab; Drug: Belimumab

INTERVENTIONS:
Drug: Rituximab — Rituximab weekly until B%<0.5% or B#<20×10^6/L
Drug: Belimumab — Belimumab every four weeks

SUMMARY:
The goal of this clinical trial is to explore the effectiveness of sequential use of rituximab and belimumab in the treatment of resistant primary juvenile Sjogren's syndrome.

Does sequential use of rituximab and belimumab reduce the activity of SS in resistant patients

Researchers will compare the disease activity before and after the treatment of sequential use of rituximab and belimumab to see if the therapy works to treat SS.

Participants will:

Recieve Rituximab each week for 2-4 times until B%<0.5% or B#<20×10^6/L Recieve Belimumab 4 weeks after the last use of Rituximab, and then every 4 weeks until week 28

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-18 years old.
2. Meets SS diagnostic AECG criteria or Japan criteria.
3. classification for "resistant patients": Application of two or more immunosuppressants or prednisone +immunosuppressive therapy for more than 3 months. One of the following conditions still exists: a) systemic involvement: polyarthritis, vasculitis, autoimmune cytopenia or involvement of skin, kidney, lung, nerve, and liver. b) constituted B cell activation: elevated IgG, light chain, high β 2MG, C4 decrease, cryoglobulinemia, monoclonal antibody c) sustained increased inflammatory markers, such as ESR
4. Agree to receive the treatment of rituximab combined with belimumab

Exclusion Criteria:

1. Previously treated with rituximab within six months, or previously treated with other biologics, including belimumab or Telitacicept
2. Participate in other clinical trials within 6 months
3. eGFR<30ml/min
4. Active infections, including but not limited to: -- Current or past infection with hepatitis B or C as defined by: Hepatitis B surface antigen positive. Hepatitis B surface antibody positive and hepatitis B core antibody positive. Hepatitis C antibody positive. -- Historically positive HIV test or test positive at screening for HIV. -- Active tuberculosis.
5. Infection history: -- Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria) -- Hospitalisation for treatment of infection within 60 days of Day 0. -- Use of parenteral (intravenous or intramuscular) antibiotics (anti-bacterials, antivirals, anti-fungals or anti-parasitic agents) within 30 days of Day 0. -- Receipt of a live-attenuated vaccine within 3 months of Day 0. -- In the investigator's opinion, participants that are at high risk for infection (including but not limited to in dwelling catheter, dysphagia with aspiration, decubitus ulcer, history of prior aspiration pneumonia or recurrent severe urinary tract infection).
6. Primary immunodeficiency
7. History of malignant neoplasm
8. Severe, progressive or uncontrolled renal, hepatic, haematological, gastrointestinal, pulmonary, cardiac or neurological disease or, in the investigator's opinion, any other concomitant medical condition or significant abnormal laboratory value that places the participant at risk by participating in this trial with the exception of diseases or conditions related to active SS
9. Comorbidities not SS related currently requiring systemic corticosteroid therapy.
10. Within 10 days before the first administration of Belimumab, IgG<4g/L or IgA<0.1g/L
11. WBC<1.5 × 109/L within 10 days before the first administration of Belimumab or neutrophils<1 × 109/L

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Respondence rate | Week 28
  In the context of the aforementioned criteria, a response is defined as the alteration of more than three of the following five indicators: a) Improvement of physician global assessment score by ≥30% b) Decrease in erythrocyte sedimentation rate (ESR) by ≥30% or normalization c) Improvement of B cell activation markers (IgG, RF) by ≥25% d) Improvement of lacrimal gland function: Improvement of Schirmer test by ≥5mm e) Improvement of salivary gland function: Increase in salivary flow rate by 25% or decrease in ultrasound score by ≥25%.

SECONDARY OUTCOMES:
Change From Baseline in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) at Week 28 | week 0 and 28
  The ESSDAI is a physician-administered tool designed to measure disease activity. It consists of 12 organ-specific 'domains' contributing to disease activity associated with the participant's Sjogren's Syndrome only (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. Overall score (ranges from 0 (no activity) to 123 (worst activity)) is calculated as sum of all individual weighted domain scores. A negative change from baseline value indicates improvement.
Change From Baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) at Week 28 | week 0 and 28
  The ESSPRI is a participant-reported questionnaire to assess subjective participant symptoms and includes 3 domains (dryness, pain, and fatigue). Each domain is scored on scale of 0-10 (0 = no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10. A negative change from baseline value indicates improvement.
the Sjögren's Tool for Assessing Response (STAR) | week 28
  The STAR is a composite responder index that includes 5 items, and the score is from 0 to 9, while more than 5 points means improvement.
Schirmer test | Week 0 and 28
  Schirmer test is a assay to detect the production of tears and less than 5mm means abnormal.
salivary flow rate | week 0 and 28
  Salivary flow rate is measured by unstimulated whole saliva. A higher salivary flow rate represents lower disease activity.
Score of salivary ultrasounds | week 0 and 28
  The Hocevar scoring system was used investigating (1) parenchymal echogenicity compared with the thyroid gland, graded 0-1; (2) homogeneity, graded 0-3; (3) presence of hypoechogenicareas, graded 0-3; (4) hyperechogenic reflections, graded 0-3 in parotid glands and 0-1 in submandibular glands; and (5) clearness of the salivary gland border, graded 0-3, in both parotid and submandibular salivary glands. Total ultrasound score was the sum of these five domains and can range from 0 to 48. A higher score usually represents more severe disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China